CLINICAL TRIAL: NCT06021977
Title: A Phase II, Single Center, Open-label Trial to Determine the Safety and Efficacy of Zanubrutinib in Refractory/Relapsed Autoimmune Hemolytic
Brief Title: The Safety and Efficacy of Zanubrutinib in Refractory/Relapsed Autoimmune Hemolytic Anemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Fang Liwei, Principal Investigator of Regenerative Medical Center, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IHBDH-IIT20230711
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Refractory/Relapsed Autoimmune Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib (Experimental): Each recruited subject will accept Zanubrutinib treatment.
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib was specifically designed to deliver complete and sustained inhibition of the BTK protein by optimizing bioavailability, half-life, and selectivity.

SUMMARY:
The sample size of this study is calculated based on Simon's two-stage design. The first stage of the study enrolled a cohort of 12 patients. If after 12 weeks at least 6 patients achieved a response, then enrollment was expanded to a total of 26 patients. The null hypothesis was unaccepted if more than 14 of 26 patients achieved the response. Accounting for a 20% dropout rate, the estimated final sample size was 33 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age from 6 to 70
* Diagnosis of Coombs-negative AIHA
* Diagnosis of warm AIHA, mixed AIHA or Evans syndrome.
* Meets the criteria of relapsed / refractory AIHA
* ECOG ≤ 3
* Willing and able to comply with the requirements for this study and written informed consent.

Exclusion Criteria:

* Diagnosis of any of the following diseases: Cold agglutinin disease, cold agglutinin syndrome, mixed AIHA, paroxysmal cold hemoglobinuria (PCH).
* Diagnosis of active stage of connective tissue disease.
* History of lymphoproliferative tumors or any other malignant.
* Diagnosis of other inherited or acquired hemolytic diseases.
* Secondary AIHA caused by drugs or infection.
* Previously received organ or stem cell transplantation.
* History of thrombosis or organ infarction.
* Received rituximab within 8 weeks before enrollment.
* Previously treated with BTK inhibitor ≥ 2 weeks.
* Received low-molecular-weight heparin or warfarin within 1 week before enrollment and need to continue the drug treatment.
* Received CYP3A4 Enzyme Inhibitors or Inducers within 1 week before enrollment and need to continue the drug treatment.
* Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment), known human immunodeficiency virus (HIV), known evidence of active infectious hepatitis B, and/or known evidence of active hepatitis C.
* Any severe and/or uncontrolled medical conditions: refractory hypertension, clinically significant cardiac diseases, renal diseases, liver diseases and metabolic diseases, etc.
* History of mental illness.
* Participation in another clinical trial within 4 weeks before the start of this trial.
* Pregnant or breast-feeding patients.
* Patients considered ineligible for the study by the investigator for reasons other than the above.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | within 12 weeks
  The percentage of patients achieved complete response, complete response with incomplete hemolysis recovery, and partial response.

SECONDARY OUTCOMES:
Incidence of adverse events and severe adverse events | within 24 weeks
Relapse free survival rate | within 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Fang, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Regenerative Medicine Center, Tianjin, Tianjin Municipality, China